CLINICAL TRIAL: NCT07062666
Title: A Multicentre Clinical Study of Near Infrared Functional Brain Imaging Combined With Eye Tracking Technique for the Auxiliary Diagnosis and Treatment Effect Prediction of Depression
Brief Title: A Multicentre Clinical Study
Status: Not yet recruiting | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Yonggui Yuan, Chairman of Scientific Committee, Zhongda Hospital
Other Study IDs: MR-32-25-015243
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: the Objective Diagnosis of Depression
MeSH Terms: interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- depressive patients
  Interventions: Drug: SSRIs; Device: fNIRS
- controls
  Interventions: Device: fNIRS

INTERVENTIONS:
Drug: SSRIs — take SSRIs for 2 weeks
  Groups: depressive patients
Device: fNIRS — All subjects receive fNIRS examination.

SUMMARY:
This study intends to conduct a multi-center, large-sample clinical trial, aiming at using multi-channel near-infrared spectroscopy to detect the characteristics of brain Oxy-Hb changes over time during cognitive activation in patients with depression before treatment and in the gender - and age-matched control group, and using eye tracking technology to detect the eye movement characteristics of patients with depression before treatment and in the gender - and age-matched control group. The sensitivity and specificity of fNIRS spectrum and eye movement index in objective diagnosis of patients with depressive disorder were calculated, and according to the HAMD reduction rate, depression patients after 2 weeks of treatment were divided into remission group and non-remission group. fNIRS imaging and eye movement indexes in depression group and normal control group were compared, fNIRS imaging and eye movement indexes in depression remission group before and after treatment, fNIRS imaging and eye movement indexes in depression remission group and non-remission group were compared at baseline to verify the biomarkers of fNIRS spectrum and eye movement indexes in predicting antidepressant efficacy. Finally, it provides reliable scientific evidence for the important role of fNIRS imaging and eye tracking technology in the diagnosis and treatment of depression.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60 years old; ② Right-handed; ③ Meet the DSM-5 diagnostic criteria for depression; ④ The current course of disease (last onset) is at least 2 weeks; ⑤HAMD-17 score ≥17 points; ⑥ No electroconvulsive therapy was received in the first six months.

Exclusion Criteria:

* A combination of another mental illness; A history of alcohol/drug dependence or smoking > 10 cigarettes/day; ③ Serious physical diseases of the heart, liver, kidney, brain and hematopoietic system, central nervous system infection, head injury, epilepsy, multiple sclerosis, toxic metabolic diseases, Parkinson's disease or intracranial tumors; ④ Family history of hereditary diseases; ⑤Endocrine system diseases such as diabetes, hyperthyroidism or hypothyroidism; ⑥ Pregnant, lactating women or photosensitivities.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: depressive patients
Sampling Method: Probability Sample
Enrollment: 2250 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
fNIRS | 2024～2025
  Sensitivity and specificity

IPD SHARING:
Plan to Share IPD: Undecided